CLINICAL TRIAL: NCT07299526
Title: Mental Health Difficulties Among Police Officers. Practices of Occupational Health Physicians and Nurses for Identifying and Referring Them to Specialized Care in France
Brief Title: Police Officers' Mental Health and Occupational Health Monitoring
Acronym: PAST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9377
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mental Health Disorder
Keywords: Mental Health Disorder; Police officers; Occupational Health
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Police officers are subject to various occupational risk factors that can contribute to the development of mental health difficulties such as depression, anxiety, and post-traumatic stress disorder. A previous study observed a low rate of access to specialized care services. Furthermore, carrying a firearm can facilitate acts of self-harm.

ELIGIBILITY:
Inclusion Criteria:

* Be an occupational physician or occupational health nurse and work with a team of national police officers,
* Agree to participate in the study,

Exclusion Criteria:

* Have been employed by the Ministry of the Interior for less than 6 months

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Occupational physician or occupational health nurse and work with a team of national police officers,
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Description of the practices of occupational health physicians and nurses | Up to 1 year
  Description of the practices of occupational health physicians and nurses involved in identifying and referring National Police officers experiencing mental health difficulties to appropriate care.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pathologie Professionnelle - Médecine du Travail - Hôpitaux Universitaires de Strasbourg, Strasbourg, France